CLINICAL TRIAL: NCT01916642
Title: Can Intravenous Lidocaine Decrease the Minimal Inducing Dose of Etomidate?: A Randomized Placebo-controlled Dose-response Study.
Brief Title: A Dose-response Study of Lidocaine and Etomidate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Niharika Dhakal, Resident,Department of Anesthesiology, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1.1
Record Dates: First submitted 2013-07-23; First posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Etomidate Overdose of Undetermined Intent
Keywords: iv lidocaine; inducing dose; etomidate; dose response
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control (Placebo Comparator): 0.9% Normal Saline is given instead of Lidocaine in the same volume and duration. Then, Etomidate 2mg intravenously every 15 seconds is given until the complete loss of consciousness as detected as the complete loss of eyelash reflex.
- Lidocaine 1mg/kg (Active Comparator): Lidocaine 1mg/kg is given intravenously within 2 minutes. Then, Etomidate 2mg intravenously every 15 seconds is given until the complete loss of consciousness as detected as the complete loss of eyelash reflex.
  Interventions: Drug: Lidocaine 1mg/kg
- Lidocaine 1.5mg/kg (Active Comparator): Lidocaine 1.5mg/kg is given intravenously within 2 minutes. Then, Etomidate 2mg intravenously every 15 seconds is given until the complete loss of consciousness as detected as the complete loss of eyelash reflex.
  Interventions: Drug: Lidocaine 1.5mg/kg
- Lidocaine 2mg/kg (Active Comparator): Lidocaine 2mg/kg is given intravenously within 2 minutes. Then, Etomidate 2mg intravenously every 15 seconds is given until the complete loss of consciousness as detected as the complete loss of eyelash reflex.
  Interventions: Drug: Lidocaine 2mg/kg
- Lidocaine 2.5mg/kg (Active Comparator): Lidocaine 2.5mg/kg is given intravenously within 2 minutes. Then, Etomidate 2mg intravenously every 15 seconds is given until the complete loss of consciousness as detected as the complete loss of eyelash reflex.
  Interventions: Drug: Lidocaine 2.5mg/kg

INTERVENTIONS:
Drug: Lidocaine 1mg/kg — The total dosage of Etomidate needed for induction of anesthesia is recorded at last.
  Other Names: Lidocaine; serial number:1303E11; Etomidate-Lipuro; serial number:11215033
  Arms: Lidocaine 1mg/kg
Drug: Lidocaine 1.5mg/kg — same as other
  Other Names: Lidocaine; serial number:1303E11; Etomidate-Lipuro; serial number:11215033
  Arms: Lidocaine 1.5mg/kg
Drug: Lidocaine 2mg/kg — same as other
  Other Names: Lidocaine; serial number:1303E11; Etomidate-Lipuro; serial number:11215033
  Arms: Lidocaine 2mg/kg
Drug: Lidocaine 2.5mg/kg — same as other
  Other Names: Lidocaine; serial number:1303E11; Etomidate-Lipuro; serial number:11215033
  Arms: Lidocaine 2.5mg/kg

SUMMARY:
IV lidocaine administration can reduce the minimal amount of Etomidate and time for induction of anesthesia.

DETAILED DESCRIPTION:
The study was carried out in West China Hospital of Sichuan University, Chengdu, China. All the patients were informed in detail about the procedure and the medications they are going to get. Patients are well informed about the beneficial and possible hazards of the medicines and procedure. Patients are also informed that they can withdraw from the study at any time if they find it uncomfortable or harmful for them. Patients' written informed consent was obtained and registered for the permission from the Hospital's Ethics Board.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for Elective Surgery,
2. age limit within 18-70 years,
3. American Society of Anaesthesiologists physical status classification I-II

Exclusion Criteria:

1. Adrenal Cortex disorder,
2. Neurologic disease,
3. Psychiatric disorders,
4. Allergic to Local anesthetic drugs,
5. Patients who have received sedatives,analgesics or opioids within the previous 24 hrs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
changes in blood pressure and heart rate. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Liu Jin, MD, Study Director — West China Hospital